CLINICAL TRIAL: NCT04070911
Title: The Effect of Oral Water and Ice Popsicle on Management of Thirst in the Immediate Postoperative Period.
Brief Title: Management of Thirst, Nursing Care, Postoperative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra eren, ASSISTANT PROFESSOR, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 55323
Record Dates: First submitted 2019-05-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Care; Nursing Caries
Keywords: Perioperative nursing; Postanesthesia care; Thirst; Water; Ice
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CONTROLLED STUDY GROUP
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients in the water group (Experimental): water group: Patients in the water group were performed oral water after their accession to PACU.
  Interventions: Other: WATER
- patients in the ice group (Experimental): ice group, Patients in the ice group were performed oral ice popsicle after their accession to PACU.
  Interventions: Other: ICE APPLICATION
- no intervention group (No Intervention): control group, the control group patients have performed rutin treatment and care without any other intervention

INTERVENTIONS:
Other: WATER — ORAL WATER
  Arms: patients in the water group
Other: ICE APPLICATION — ICE APPLICATION
  Arms: patients in the ice group

SUMMARY:
The study was conducted to determine the effect of oral water and ice popsicle on management of thirst in the immediate postoperative period as experimental.

DETAILED DESCRIPTION:
Also, it is aimed to evaluate validity and reliability of "Safety Protocol for Management Thirst in the Immediate Postoperative Period Protocol" which is used to take oral water and ice of patients in the immediate postoperative period, as administrative. The study was conducted with 150 patients who are transferred to the postanesthesia care unit (PACU) after their operation and met study criteria. Patients divided into three groups as the study (water group=50, ice group=50) and control (n=50). Patients in the study group were performed oral water/ice popsicle after their accession to PACU. However, the control group patients have performed rutin treatment and care without any other intervention. Physiologic variables and symptoms with thirst were followed in every three group patients at certain times. Data were evaluated by using NCSS (Number Cruncher Statistical System) 2007 program.

ELIGIBILITY:
Inclusion Criteria:

1. have a surgical operation other than gastrointestinal system surgery,
2. Surgical fasting duration is at least 8 hours,
3. According to the American Society of Anesthesiologists (ASA) classification; Class I, II and III;
4. Having the ability to express the thirst status verbally and experiencing moderate or severe thirst when the thirst status is evaluated by VAS,
5. The duration of anesthesia is longer than 1 hour and accepted into the PACU after surgery.

Exclusion Criteria:

1. have a second surgical intervention during hospitalization,
2. The need of intensive care after surgery,
3. Having problems in the process of separation from respiratory support after surgical intervention,
4. A change in the state of consciousness after surgical intervention / acute confusion,
5. Liquid electrolyte imbalance,
6. Patients with difficulty in swallowing or restriction of oral fluid intake,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
THIRSTY SCALE | first 30 minutes after the surgery
  Thirsty and symptoms of thırsty evaluated via vısual analog scale which containing numbers from zero to ten (0-10), "0" is the minumun point, "10" is the maximum point, higher values represent a better situation.

SECONDARY OUTCOMES:
The blood pressure measurements in the first 30 minutes after surgery | first 30 minutes after surgery
  Blood pressure was obtained from the monitor data of patients who were monitored postoperatively. Blood pressure was measured as "mmHg".
The heart rate measurements in the first 30 minutes after surgery | first 30 minutes after surgery
  Heart rate was obtained from the monitor data of patients who were monitored postoperatively. heart rate refers to the number of beats per minute.
The respiratory rate measurements in the first 30 minutes after surgery | first 30 minutes after surgery
  The respiratory rate was obtained from the monitor data of the patients who were monitored postoperatively. respiration rate is the sum of inspiration and expiration per minute.
The body temperature measurements in the first 30 minutes after surgery | first 30 minutes after surgery
  Body temperature was obtained from the monitor data of patients who were monitored postoperatively. body temperature was recorded with the degree system in degrees Celsius.

CONTACTS AND LOCATIONS:
Overall Officials: seher deniz öztekin, Prof.Dr., Study Director — thesis advisor
Locations (1):
- Istanbul Medipol University, Kavacık, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT04070911/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT04070911/SAP_001.pdf